CLINICAL TRIAL: NCT00982514
Title: Thromboembolic Complications Related to Asparaginase in Children With ALL Treated According to NOPHO ALL 2008
Brief Title: Thromboembolic Complications Related to Asparaginase in Children With Acute Lymphoblastic Leukemia (ALL) Treated According to NOPHO ALL 2008
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ASP NOPHO 2008
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Thromboembolism; Acute Lymphoblastic Leukemia
Keywords: Asparaginase; thrombosis; ALL; central line
MeSH Terms: conditions — Thromboembolism; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard dose asparaginase: Children who according to the protocol NOPHO ALL 2008 receive standard dose asparaginase
- Reduced dose asparaginase: Children who receive reduced dose asparaginase according to NOPHO ALL 2008

SUMMARY:
The study will examine the prevalence of venous thromboembolism in children with acute lymphoblastic leukaemia treated in accordance with NOPHO ALL-2008. The investigators will prospectively study clinical symptomatic thromboses, asymptomatic central line-associated thromboses, and infections.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukaemia,
* Age 1 year to 16 years old,
* Central line,
* Protocol NOPHO ALL 2008.

Exclusion Criteria:

* Refusal of participation,
* Treated according to protocol other than NOPHO ALL 2008.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Oslo University Hospital, Department of Pediatrics
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Clinical evident thrombosis | 33 weeks
Asymptomatic central line-associated thrombosis | 33 weeks

SECONDARY OUTCOMES:
Positive blood culture | 33 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Ruud, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet, Dep of Pediatrics, Oslo, Oslo County, Norway